CLINICAL TRIAL: NCT00322517
Title: A Phase 2 Study Of The Efficacy And Safety Of SU-014813 In Patients With Metastatic Breast Cancer
Brief Title: Study Of The Efficacy And Safety Of SU-014813 In Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6191007
Record Dates: First submitted 2006-04-17; First posted 2006-05-08 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SU014813 (Experimental)
  Interventions: Drug: SU014813

INTERVENTIONS:
Drug: SU014813 — 100 mg capsule/day for 6 cycle of 21 days

SUMMARY:
To determine the antitumor efficacy and the safety of SU-014813 at a dose of 100 mg orally once daily in patients with Metastatic Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of metastatic breast adenocarcinoma that is not amenable to surgery, radiation, or combined modality therapy with curative intent.
* Must have received prior treatment with an anthracycline and a taxane either concurrently or sequentially in the adjuvant and/or advanced disease treatment settings. Patients may have received as many as 2 other chemotherapy regimens in the advanced disease setting. Patients whose tumors are Her-2-positive must have received prior trastuzumab therapy. Prior hormonal therapy or immunotherapy in the adjuvant and/or advanced/metastatic disease settings is permitted. Prior treatment with surgery, radiotherapy, chemoembolization therapy, or cryotherapy is allowed if these therapies did not affect the areas of measurable disease.

Exclusion Criteria:

* Prior treatment with >/= 3 regimens of chemotherapy in the metastatic disease setting beyond those containing anthracyclines and taxanes
* Uncontrolled brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients should have completed surgery or radiation therapy for existing brain metastases, should not have documented increase in size over the previous 3 months and should be asymptomatic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the antitumor efficacy of single agent SU-014813 at a dose of 100 mg orally once daily in patients with MBC | June 2008

SECONDARY OUTCOMES:
To assess onset and duration of tumor control and 1-year survival rate | AUG 2008
To evaluate the safety of SU-014813To assess patient reported outcomes | AUG 2008
To determine SU-014813 plasma trough concentration (Ctrough) | AUG 2008
To explore the relationship between Ctrough and efficacy, safety, and biomarkers | AUG 2008
To explore the correlations of cancer biomarkers with treatment-related outcomes | AUG 2008

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (7):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Valancia, California
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Memphis, Tennessee
- Germany (3):
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Magdeburg
  - Pfizer Investigational Site, Marburg
- Italy (4):
  - Pfizer Investigational Site, Chieti Scalo
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Mirano (VE)
  - Pfizer Investigational Site, Udine
- Netherlands (2):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Rotterdam
- United Kingdom (4):
  - Pfizer Investigational Site, Manchester, M20 4bx
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6191007&StudyName=Study%20Of%20The%20Efficacy%20And%20Safety%20Of%20SU-014813%20In%20Patients%20With%20Metastatic%20Breast%20Cancer%0A